CLINICAL TRIAL: NCT05158361
Title: Effectiveness and Safety of Acupuncture for Overactive Bladder in Adults: A Random Control Clinical Trial
Brief Title: Acupuncture for Overactive Bladder in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Ran Pang, Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019S443
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Acupuncture
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Participants will receive acupuncture.
  Interventions: Other: Acupuncture
- Sham acupuncture (Sham Comparator): Participants will receive sham acupuncture.
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Acupuncture — Participants will receive acupuncture, three times per week for eight weeks. The selected acupoints include bilateral BL33, BL35, SP6, and ST36. All acupoints areas have been sterilized before acupuncture. For BL33, a needle (Ф0.40×100mm) will be inserted with an angle of 60° in an inferomedial direction at a depth of 90-100mm. For BL35, the same needle will be inserted with a direction to the ischial rectal fossa at a depth of 60-70 mm deep. For SP6 and ST36, needles (Ф0.30×50mm) will be directly inserted at a depth of 25-30 mm deep. After the needles are inserted, a portable electro-acupuncture machine will be connected to the handles of needles located in BL33 and BL35 to provide the electrical stimulation for 30 minutes with a disperse-dense wave (4/20Hz). All current intensities will be as high as can be tolerated.
  Arms: Acupuncture
Other: Sham acupuncture — The sham acupoints will be located at 20 mm outward to BL33, BL35, SP6, and ST36, and the needless will be inserted with a depth of 2 mm. The BL33 and BL35 will not receive any electrical stimulation, though the handles of needles will be connected to the same machine as the acupuncture group, and the parameter setting and course are also the same.
  Arms: Sham acupuncture

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of acupuncture for treating overactive bladder in adults.

DETAILED DESCRIPTION:
This randomized, controlled trial is aimed to assess the effectiveness and safety of acupuncture in the treatment of overactive bladder (OAB) in adults. Eligible participants will be randomly allocated to acupuncture or sham acupuncture.

To minimize the evaluation bias, the outcome assessors and statisticians will be masked to treatment allocation besides participants.

ELIGIBILITY:
Inclusion Criteria:

* Present symptoms of urinary frequency and urgency for more than 3 months.
* With a total score of more than 3 points on the overactive Bladder Symptom Score (OABSS) and a score of more than 2 points on question 3 of OABSS.

Exclusion Criteria:

* With other lower urinary tract disorders (e.g. urinary tract infection, bladder outlet obstruction, neurogenic bladder, interstitial cystitis, etc.)
* With previous pelvic floor surgery or a post-void residual urine volume more than 100 mL.
* With neurological disease or psychiatric illness.
* Taking medications affecting lower urinary tract function.
* With contraindications to acupuncture.
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in number of micturition episodes per 24 hours | Before treatment (baseline), 8 week (post-treatment) and 12 week (follow-up)
  Assessed by 72 h bladder diary

SECONDARY OUTCOMES:
Number of urinary urgency episodes per 24 hours | Before treatment (baseline), 8 week (post-treatment) and 12 week (follow-up)
  Assessed by 72 h bladder diary
Number of daytime micturition episodes per 24 hours | Before treatment (baseline), 8 week (post-treatment) and 12 week (follow-up)
  Assessed by 72 h bladder diary
Number of nocturia episodes per 24 hours | Before treatment (baseline), 8 week (post-treatment) and 12 week (follow-up)
  Assessed by 72 h bladder diary
Change in mean volume voided per micturition | Before treatment (baseline), 8 week (post-treatment) and 12 week (follow-up)
  Assessed by 72 h bladder diary
Change in OABSS questionnaire | Before treatment (baseline), 8 week (post-treatment) and 12 week (follow-up)
  Assessed by Overactive Bladder Symptom Score (OABSS) questionnaire. OABSS includes 4 questions about individual symptoms, and the total score ranged from 0 to 15, with higher scores indicating more severe symptoms. The minimal important difference (MID) for the OABSS is 3 points.
Change in OAB-q SF questionnaire | Before treatment (baseline), 8 week (post-treatment) and 12 week (follow-up)
  Assessed by overactive bladder questionnaire short form (OAB-q SF) questionnaire. OAB-q SF includes 6 questions on 6-point Likert-type scales, with the outcomes transformed to a 0-100 point scale in which higher scores indicate more severe symptoms. The minimal important difference (MID) for the OAB-q SF is 11 points.
Urinary NGF/Cr level | Before treatment (baseline), 8 week (post-treatment)
  Measured by human nerve growth factor (NGF) ELISA Kit. NGF/Cr: NGF normalized to urine creatinine (Cr)
Urinary BDNF/Cr level | Before treatment (baseline), 8 week (post-treatment)
  Measured by human brain derived neurotrophic factor (BDNF) ELISA Kit. BDNF/Cr: BDNF normalized to urine creatinine (Cr)
Urinary MCP-1/Cr level | Before treatment (baseline), 8 week (post-treatment)
  Measured by human monocyte chemoattractant protein-1 (MCP-1) ELISA Kit. MCP-1/Cr: MCP-1 normalized to urine creatinine (Cr)

CONTACTS AND LOCATIONS:
Overall Officials: Ran Pang, MD, Principal Investigator — Guang'anmen hospital
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The agreement for sharing IPD is not designed to be signed in informed consent form.

REFERENCES:
- [Derived] Hargreaves E, Baker K, Barry G, Harding C, Zhang Y, Kandala NB, Zhang X, Kernohan A, Clarkson CE. Acupuncture for treating overactive bladder in adults. Cochrane Database Syst Rev. 2022 Sep 23;9(9):CD013519. doi: 10.1002/14651858.CD013519.pub2. PMID 36148895